CLINICAL TRIAL: NCT01860807
Title: Randomized Trial of Ibudilast for Methamphetamine Dependence
Brief Title: Trial of Ibudilast for Methamphetamine Dependence
Acronym: IBUD ph II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Keith Heinzerling, Associate Professor in Residence, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1R01DA035054-01 (NIH); R01DA035054 (NIH)
Record Dates: First submitted 2013-05-20; First posted 2013-05-23 (Estimated); Results first posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Methamphetamine Dependence; HIV Infection
Keywords: methamphetamine; ibudilast; HIV
MeSH Terms: conditions — HIV Infections | interventions — ibudilast

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ibudilast (Experimental): Ibudilast 50 mg twice daily
  Interventions: Drug: Ibudilast
- Placebo (Placebo Comparator): matching placebo twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibudilast
  Arms: Ibudilast
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective of this study is to test the safety and potential efficacy of ibudilast to treat methamphetamine dependence. The study hypotheses are that ibudilast will reduce methamphetamine use and increase treatment retention more than placebo among patients seeking treatment for methamphetamine dependence. As HIV infection is a common complication of methamphetamine dependence, half of the participants will be HIV positive and the study will assess whether ibudilast also improves HIV related outcomes (e.g. medication adherence, CD4 count, risk behaviors).

DETAILED DESCRIPTION:
Ibudilast (IBUD) is a macrophage migration inhibitory factor (MIF) and phosphodiesterase (PDE)-4 and -10 inhibitor at peak clinical exposures (Rolan, Hutchinson et al. 2009) that increases glial cell line-derived neurotrophic factor (GDNF) expression (Mizuno, Kurotani et al. 2004) and reduces microglial activation (Suzumura, Ito et al. 1999; Suzumura, Ito et al. 2003), including HIV-induced glial activation (Kiebala and Maggirwar 2011). IBUD significantly reduces methamphetamine (MA) prime- and stress-induced reinstatement of MA seeking in rats (Beardsley, Shelton et al. 2010) and has multiple effects that may make it an effective treatment for MA dependence including amelioration of dopaminergic and neuroinflammatory dysfunction. Multiple studies implicate glial cells in a variety of neurodegenerative diseases (Hirsch and Hunot 2009; Sidoryk-Wegrzynowicz, Wegrzynowicz et al. 2011) including MA dependence and HIV infection (Nath 2010). Activated glial cells secrete pro-inflammatory mediators (Minghetti, Ajmone-Cat et al. 2005) that may exacerbate MA-induced dopaminergic dysfunction. Glial cells also produce neurotrophic factors, including GDNF, which may ameliorate dopaminergic dysfunction (Pascual, Hidalgo-Figueroa et al. 2008). Thus, IBUD may be an effective medication for MA dependence due to its modulation of glial cell activation resulting in amelioration of dopaminergic and neurocognitive dysfunction and improved treatment outcomes in MA dependence. IBUD may also have unique effects in HIV positive MA users as it may additionally block the degradation of neuronal integrity seen in HIV infection (Chana, Everall et al. 2006; Dash, Gorantla et al. 2011).

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older;
2. meet DSM-IV-TR criteria for MA dependence (SCID verified);
3. a MA-positive urine drug screen at one or more visit during the two week lead-in period;
4. seeking treatment for MA problems;
5. willing and able to comply with study procedures;
6. provide written informed consent;
7. English speaking
8. reside within 35 miles of the clinical research site; and
9. if female of childbearing potential, not pregnant or lactating and willing to use a medically reliable method of birth control during the trial (e.g., birth control pills, Depo-Provera, and/or condoms with spermicide).

Exclusion Criteria:

1. a medical condition that, in the study physician's judgment, may interfere with safe study participation (e.g., active TB; unstable cardiac, renal, or liver disease; uncontrolled hypertension; unstable diabetes);
2. CD4 count < 50 cells/mm3 (suggestive of advanced HIV infection)
3. AST, ALT, or GGT > 3 times upper normal limit;
4. A corrected QT of > 450 msecs in men or > 460 msec in women on at least two ECGs during the baseline period, or clinical risk factors for Torsades de Pointes (e.g. (e.g., heart failure, hypokalemia, family history of Long QT Syndrome), or requiring ongoing treatment with concomitant medication(s) with established risk of Torsades de Pointes (e.g. Amiodarone, Arsenic trioxide, Astemizole, Bepridil, Chloroquine, Chlorpromazine, Cisapride, Citalopram, Clarithromycin, Disopyramide, Dofetilide, Domperidone, Droperidol, Erythromycin, Flecainide, Halofantrine, Haloperidol, Ibutilide, Levomethadyl, Mesoridazine, Methadone, Moxifloxacin, Pentamidine, Pimozide, Probucol, Procainamide, Quinidine, Sotalol, Sparfloxacin, Terfenadine, Thioridazine, Vandetanib);
5. current ongoing treatment with psychotropic medications (e.g., antidepressants, antipsychotics, antiepileptics, sedative/hypnotics, narcotic analgesics);
6. a neurological disorder (e.g., organic brain disease, dementia) or a medical condition which would make study agent compliance difficult or which would compromise informed consent;
7. a major psychiatric disorder not due to substance abuse (e.g., schizophrenia, bipolar disorder) as assessed by the SCID;
8. attempted suicide in the past 3 years and/or serious suicidal intention or plan in the past year as assessed by the C-SSRS;
9. currently on prescription medication that is contraindicated for use with IBUD including alpha or beta agonists, theophylline, or other sympathomimetics;
10. current dependence on cocaine, opiates, alcohol, or benzodiazepines as defined by DSM-IV-TR;
11. alcohol dependence within the past year;
12. greater than one urine specimens during the lead-in with a riboflavin concentration of < 900 ng/ml as assessed via UV fluorescence;
13. a history of sensitivity to IBUD; or
14. any other circumstances that, in the opinion of the investigators, would compromise participant safety;
15. current participation in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2013-07; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Heinzerling, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Vine Street Clinic, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ibudilast: Ibudilast 50 mg twice daily
  Ibudilast
- Placebo: matching placebo twice daily
  Placebo
Period: Overall Study
Arm/Group | Ibudilast | Placebo
Started | 64 | 61
Completed | 34 | 32
Not Completed | 30 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibudilast | Placebo | Total
Number analyzed (Participants) | 64 | 61 | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (9.0) | 42.8 (10.5) | 41.9 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 18 | 33
  Male | 49 | 43 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 30 | 60
  Not Hispanic or Latino | 34 | 31 | 65
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 7 | 7 | 14
  White | 29 | 30 | 59
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 21 | 19 | 40
Baseline methamphetamine use on 26 or more days per month [Count of Participants; unit: Participants] | 33 | 33 | 66

OUTCOME MEASURES:

1. Primary Outcome: Methamphetamine Use
Description: End of treatment methamphetamine abstinence
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Ibudilast | Placebo
Number analyzed (Participants) | 64 | 61
Participants | 9 | 10

ADVERSE EVENTS:
Time Frame: 12 week medication treatment period and 4 week post-treatment follow-up period
Arm/Group | Ibudilast | Placebo
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/61
Serious Adverse Events (participants affected / at risk) | 2/64 | 1/61
Other Adverse Events (participants affected / at risk) | 57/64 | 32/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibudilast (N=64) | Placebo (N=61)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1)
Suicide Attempt (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ibudilast (N=64) | Placebo (N=61)
Headache (Nervous system disorders) | 32 | 11
Nausea (Gastrointestinal disorders) | 11 | 9
Insomnia (Psychiatric disorders) | 10 | 5
Diarrhea (Gastrointestinal disorders) | 8 | 7

LIMITATIONS AND CAVEATS:
Study did not determine if ibudilast may help patients who have stopped methamphetamine use prior to starting medication

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-11): https://cdn.clinicaltrials.gov/large-docs/07/NCT01860807/Prot_SAP_000.pdf